CLINICAL TRIAL: NCT00350363
Title: One Hour Preoperative Gatifloxacin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Ta, PI, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 5004
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Ophthalmic Surgery
MeSH Terms: interventions — Gatifloxacin

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- 1 hour gatifloxacin (Active Comparator): presence of conjunctival bacteria 1 hour after administration of topical gatifloxacin
  Interventions: Drug: Zymar

INTERVENTIONS:
Drug: Zymar — zymar qid
  Other Names: gatifloxacin

SUMMARY:
Comparison of 1 day versus 1 hour application of topical Zymar.

ELIGIBILITY:
Inclusion Criteria:

* ophthalmic surgery

Exclusion Criteria:

* taken antibiotics, allergic to fluoroquinolones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ta, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Day of Gatifloxacin: eyes receiving gatifloxacin 4 times per day 1 day before surgery
Period: Overall Study
Arm/Group | 1 Day of Gatifloxacin
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: patients undergoing eye surgery
Arm/Group | 1 Day of Gatifloxacin
Number analyzed (Participants) | 60
Age, Continuous [Mean (Full Range); unit: years] | 68 [50 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Positive Culture
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | 1 Day of Gatifloxacin
Number analyzed (Participants) | 60
participants | 17

ADVERSE EVENTS:
Arm/Group | 1 Day of Gatifloxacin
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No